CLINICAL TRIAL: NCT07239726
Title: CLINICAL INVESTIGATION TO EVALUATE THE EFFICACY AND SAFETY OF EPILADY PROTOTYPE DEVICE FOLLOWED BY APPLICATION OF A TOPICAL FORMULA ON DEPIGMENTATION OF LENTIGO SPOTS IN HEALTHY WOMEN PARTICIPANTS - STUDY UNDER DERMATOLOGICAL CONTROL
Brief Title: CLINICAL INVESTIGATION TO EVALUATE THE EFFICACY AND SAFETY OF EPILADY PROTOTYPE DEVICE FOLLOWED BY APPLICATION OF A TOPICAL FORMULA ON DEPIGMENTATION OF LENTIGO SPOTS
Acronym: EPILADY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EV2409-0042 / ID 24-14993
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Solar Lentigo
Keywords: solar lentigo,; Laser treatment
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LASER (Experimental): Healthy participants aged between 35 and 70 years old with presence of at least two solar lentigo on each hand or forearm, with each spot measuring less than 100 mm x 100 mm as assessed by the investigator
  Interventions: Other: LASER
- LASER AND ACTIVE FLORMULA (Active Comparator): Healthy participants aged between 35 and 70 years old with presence of at least two solar lentigo on each hand or forearm, with each spot measuring less than 100 mm x 100 mm as assessed by the investigator
  Interventions: Combination Product: LASER AND ACTIVE FORMULA

INTERVENTIONS:
Other: LASER — Application of laser once a weeks by dermatologist on spot and application of sunscreen twice a day ( morning and midday) for 3 months
  Arms: LASER
Combination Product: LASER AND ACTIVE FORMULA — application of laser once a week by dermatologist, active formula twice a day ( morning and evening) and sunscreen formula twice a day (morning and midday) for 3 months
  Arms: LASER AND ACTIVE FLORMULA

SUMMARY:
To assess the efficacy of the Epilady investigational device, used with and without a topical depigmenting formula, in reducing the appearance of lentigo spots on the hands and forearms of healthy female participants over an 84-day period

DETAILED DESCRIPTION:
Rational The investigational product in this clinical investigation, the Epilady laser-based device, applies the principle of selective photothermolysis to target melanin within pigmented lesions. It uses diode laser technology at either 660 nm or 808 nm, selected according to the participant's skin phototype, and is equipped with a camera-guided targeting system and integrated safety sensors for precise and controlled energy delivery. The device has been classified as a Class IIb medical device in the EU, intended for the permanent reduction of pigmentation such as lentigines.

Design:

This is a prospective, open-label, randomized, intra-individual controlled clinical investigation conducted in healthy female participants aged 35 to 70 years. The clinical investigation is designed to evaluate the efficacy and safety of the Epilady prototype laser medical device, used alone or in combination with a cosmetic depigmenting formula, in reducing the pigmentation of lentigo spots on the hands and lower forearms.

Following inclusion, the left and right hands (or forearms) of each participant will be randomized:

* One side will receive weekly laser treatments with the device alone, while
* The contralateral side will receive weekly laser treatments with the device followed by twice-daily application of the cosmetic formula starting 24 hours after each laser session and continuing for the remainder of the 84-day period.

Reglementation The clinical investigation will be conducted in compliance with Good Clinical Practice (GCP) guidelines and applicable regulatory requirements for medical device investigations, ISO 14155.

Objectifs & Statistiques Safety analyses will be performed on the SS population, while efficacy analyses will be primarily performed on the ITT population. If the sample size between the PP and ITT populations differs by more than 10%, the efficacy analysis will also be performed on the PP population.

Pigmentation intensity by L'Oréal color chart:

The score of the "balance of red/yellow" will be coded as follows:

* G (red): a score of 7 will be attributed
* H: a score of 6 will be attributed
* I: a score of 5 will be attributed
* J: a score of 4 will be attributed
* K: a score of 3 will be attributed
* L: a score of 2 will be attributed
* M (yellow): a score of 1 will be attributed Thus, a decrease in the score from D0 onwards, will indicate a change of skin colour from red to yellow.

The change in red/yellow component [letters G (red tendency) to M (yellow tendency)] will be added to the change in lightness [numbers 19 (dark skin) to 5 (fair skin)] for analysis purposes, e.g. a change from G18 to J15 will correspond to a change of -6 units.

On each assessed area separately (lentigo spot and adjacent) and each side, the significance of the change from baseline will be assessed using a one sample t-test (versus 0, which would indicate no change).

The assessment of the change from baseline on each side will be assessed using a Paired Samples t-test or the Wilcoxon Signed Ranked, depending on the normality of the data. Similarly, the comparison of the two sides will be assessed using the same statistical tests. The normality of the data will be tested at 1% of the Shapiro Wilk test.

Lentigines Global Improvement Scale (LGIS):

At each visit, the comparison of the two treatments will be investigated using a Wilcoxon Signed Rank test.

Self-assessment efficacy questionnaires:

The answers to the efficacy questionnaire will be summarized in a frequency table by category, together with 100% stacked bar charts.

Safety assessment:

AEs will be listed by participants including time of onset, time from the first administration of clinical investigation drug, duration, intensity, action taken, corrective therapies, outcome, relationship to clinical investigation drug and seriousness.

Local tolerance will be reported descriptively.

For the comparison of treatments, the null and alternative hypotheses are as follows:

H0: There is no difference between the two treatments H1: There is difference between the two treatments To claim superiority of the device + cosmetic formula, the null hypothesis should be rejected, and the average score should be in favor of the device + cosmetic formula.

Significance level :The null hypothesis will generally be rejected if a p-value less than 0.05 (5% significance level) is produced by the statistical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female participants aged between 35 and 70 years old at the time of inclusion.
* All Fitzpatrick skin phototypes (I to VI) are eligible; groups I-II and V-VI should include at least one participant per group.
* Presence of at least two solar lentigo (dark spots) on each hand or forearm, with each spot measuring less than 100 mm x 100 mm as assessed by the investigator.
* Participant has read, understood, and accepted the constraints of the clinical investigation.
* Participant has provided written informed consent to participate in the clinical investigation.
* Participant is able to understand the language used in the investigational site and comprehend the information provided.
* Participants are cooperative and compliant, aware of the clinical investigation requirements and willing to adhere to the full duration of participation and follow-up visits, in line with the CIP requirements.
* Women of childbearing potential must commit to using an effective contraceptive method throughout the clinical investigation period and for at least three months prior to the inclusion visit, with no changes during that time.

Exclusion Criteria:

* • Participants with dry or sensitive skin, as assessed by the investigator.

  * Participants who have used cosmetic products with exfoliating or astringent claims on the hands within 4 weeks prior to the baseline visit.
  * Participants who have used any home-use or professional low-level laser therapy (LLLT) or have participated in clinical studies involving LLLT within the 6 months preceding the baseline visit
  * History of light-induced seizures or chronic migraine disorders.
  * History of photosensitivity or photoallergic reactions.
  * Presence of underlying dermatological conditions on the hands/forearms that, in the opinion of the investigator, could interfere with the clinical investigation assessments.
  * A family history of melanoma in first- or second-degree relatives (parents or grandparents).
  * Presence of excessive moles, non-lentigo pigmented lesions, tattoos, scars, or irritated skin in the test area that could affect the validity of the investigation.
  * History of surgical procedures involving the areas designated for treatment.
  * Participants who have been exposed to or plan to be exposed to sunbathing or artificial UV sources (e.g., mountain sports, phototherapy, tanning salons) within 1 month before the clinical investigation start or during the clinical investigation period.
  * Use of suntan or self-tanning products within the 2 weeks preceding the baseline visit.
  * Change in cosmetic habits (e.g., moisturizers, skincare, shower gels) during the 2 weeks prior to baseline.
  * Use of any medications, topical treatments, skincare products, or aesthetic procedures listed in the CIP without observing the required wash-out periods, or unwillingness/inability to comply with those restrictions during the clinical investigation.
  * Participant who cannot be contacted by telephone in case of emergency
  * Participant in an exclusion period or participating in another biomedical research clinical investigation (self-reported)
  * Intellectual/mental inability to follow clinical investigation instructions (if suspected) or incapacitation.
  * Participants working for the contract research organization (CIDP) in charge of this clinical investigation.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Change of the pigmentation intensity of solar lentigo | baseline to 3 months
  The investigator will perform a standardized clinical evaluation of the targeted lentigo lesions, grading pigmentation intensity using a standardized Color Chart (2021-EV-FR-ICE-Color Chart Procedure, see figure 2) to assess the darkness of each lentigo lesion compared to the surrounding skin.
Global tolerance | 1 month to 3 months
  The investigator will assign an overall tolerance score for the treatment area at each visit using the following scale 1: very good ; 2: good; 3: Moderate; 4: Bad

SECONDARY OUTCOMES:
Lentigines Global Improvement Scale (LGIS) | baseline to 3 months
  The investigator will assess the overall improvement of each treatment area using the Lentigines Global Improvement Scale (LGIS). This scale rates changes in pigmentation, lesion size, and skin homogeneity with 7 grades ( 0 : Completrely clear to 6 : worse)
Self assessment questionnaire | 3 months
  Participants will complete a subjective evaluation questionnaire to capture their perception of treatment outcomes.
  The questionnaire, using a 5-point scale (1 = Disagree to 5 = Agree), will include items on visible results, comfort during and after use, perceived reduction in pigmentation , improvement in overall skin appearance (tone, brightness, clarity), and overall satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- CIDP Ltée, Phoenix, Mauritius